CLINICAL TRIAL: NCT05296304
Title: A Phase Ib Trial Combining Bexarotene With Ultra-Low Dose Total Skin Electron Beam (Tseb) Radiotherapy For The Treatment Of Diffuse Cutaneous T-Cell Lymphomas
Brief Title: A Study of Bexarotene Combined With Radiotherapy in People With Mycosis Fungoides
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-501
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cutaneous T-cell Lymphoma
Keywords: Bexarotene; Radiotherapy; Mycosis Fungoides; 21-501
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides | interventions — Bexarotene

STUDY DESIGN:
Intervention Model Description: This is a Phase I, single-arm therapeutic study for patients with diffuse cutaneous T-cell lymphomas (CTCL).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bexarotene Combined With Radiotherapy (Experimental): Patients will be initiated on bexarotene 150 mg daily on Day 1, with dose increase to 300 mg daily on Day 15. Patients will receive Cycle 1 of TSEB on Day 22 (with 2 Gy given on two consecutive days -Day 22 and 23), with safety assessment on Day 52. Efficacy will first be assessed on Day 52 and then again on Day 82 by global response assessment, including mSWAT. Patients who have less than 70% reduction from baseline mSWAT score will be eligible for subsequent cycles of TSEB (administered as 4 Gy over 2 consecutive days), until mSWAT score reduction of ≥ 70%, and up to a total of 6 cycles. Treatment may continue until disease progression, unacceptable toxicity, recommended termination by treating physician, or termination of the study.
  Interventions: Drug: Bexarotene; Radiation: Total Skin Electron Beam (TSEB)

INTERVENTIONS:
Drug: Bexarotene — Orally every day starting at the dose of 150 mg/day flat dose. At Day 15, if the treatment is tolerated, patients will escalate the dose of bexarotene to 300 mg/day, and that dose will remain constant during the rest of the study.
  Other Names: Targretin®
Radiation: Total Skin Electron Beam (TSEB) — At Day 21, if the bexarotene has shown to be tolerated, patients will receive the first dose of TSEB (2 Gy x 2).

SUMMARY:
The researchers are doing this study to test the safety of combining bexarotene with TSEB radiotherapy in people who have a common form of CTCL called mycosis fungoides (MF).

Bexarotene is a form of vitamin A that activates proteins called retinoid X receptors, which may stop the growth of cancer cells and kill them. TSEB radiotherapy is a type of radiation therapy that treats the entire surface of the skin with very low doses of radiation to kill cancer cells and shrink tumors. This type of radiation does not pass through the outer layers of the skin into the tissues and organs below the skin.

The study researchers think that giving bexarotene treatment at the same time as treatment with TSEB radiotherapy may be more effective against MF than either treatment given alone or in sequence (one after the other).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Pathologically confirmed cutaneous T-cell lymphoma consistent with mycosis fungoides (MF) based on biopsy done or reviewed at MSKCC
* Stage IB or higher MF per ISCL/EORTC criteria; concurrent diagnosis of Sézary syndrome permissible. Patients who have not had prior systemic therapies and refractory/relapsed patients are eligible.
* Baseline mSWAT score of at least 10
* Stable topical steroids or systemic antipruritic agent (e.g. antihistamines, doxepin, GABA analogs) preceding study entry is permissible, but no new prescribed or over the counter topical or systemic anti-pruritics started post-enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Ability to provide informed consent

Exclusion Criteria:

* Any oral retinoid therapy for any indication within 3 weeks of the first dose of study drug
* Prior TSEB (prior focal skin-directed RT acceptable)
* Concurrent diagnosis of systemic anaplastic large cell lymphoma (ALCL) or another non-Hodgkin lymphoma
* Concurrent diagnosis of additional non-skin malignancy
* Pregnancy
* Patients unwilling to use two forms of barrier contraception while taking study medication
* Receipt of treatment with another investigational device or drug (at present or within 2 weeks of enrollment)
* Familial hypertriglyceridemia or other medical conditions in which use of bexarotene would be contraindicated
* High likelihood of protocol non-compliance (in opinion of investigator)
* Systemic steroids within two weeks of first dose of study drug (patients on systemic steroids for non-disease related conditions will be permitted per investigator discretion)

Prohibited concurrent medications

* Gemfibrozil is contraindicated as may increase bexarotene concentrations
* Bexarotene is a minor CYP3A4 substrate: avoid strong/moderate CYP3A4 inducers and inhibitors, if possible, but concomitant use is not a contraindication Bexarotene is a moderate CYP3A4 inducer: avoid concurrent administration with CYP3A4 sensitive substrates, for which minimal concentration changes may lead to therapeutic failures of the substrate (e.g. cyclosporine, tacrolimus, sirolimus, quinidine, fentanyl), if possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of radiation dermatitis grade 3+ | 1 month post-treatment
  as defined by number of patients who develop CTCAE, v. 5, grade 3+ toxicities at 1 month post-treatment.

SECONDARY OUTCOMES:
Overall skin response rate | up to 82 days post-TSEB
  For patients with mycosis fungoides without blood involvement, the response criteria will be based upon modified international consensus guidelines.26 Specifically, skin response will be assessed by the Modified Severity Weighted Assessment Tool (mSWAT). For the purposes of this protocol, overall skin response will be considered to be either CR or PR.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Imber, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm